CLINICAL TRIAL: NCT04889365
Title: The Use of SG Diagnostics COVID-19 Antigen Rapid Test Kit for Self-testing as a Method for Reduction SARS-CoV-2
Brief Title: COVID-19 Antigen Rapid Test Kit
Acronym: SETCOV
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Polish Society of Disaster Medicine (Other)
Responsible Party: Sponsor
Other Study IDs: PTMK_2021_01
Record Dates: First submitted 2021-05-10; First posted 2021-05-17 (Actual); Last update posted 2021-05-17 (Actual); Status verified 2021-05

CONDITIONS: SARS-CoV2 Infection
Keywords: SARS-CoV-2; COVID-19; symptoms; test
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- COVID-19 positive, asymptomatic: COVID-19 positive, asymptomatic (i.e. no current symptoms of COVID-19, confirmed PCR positive for COVID-19)
  Interventions: Diagnostic Test: SG Diagnostics COVID-19 Antigen Rapid Test Kit; Diagnostic Test: Polymerase chain reaction (PCR) test
- COVID-19 positive, symptomatic: COVID-19 positive, symptomatic (i.e. current symptoms of COVID-19, confirmed PCR positive for COVID-19)
  Interventions: Diagnostic Test: SG Diagnostics COVID-19 Antigen Rapid Test Kit; Diagnostic Test: Polymerase chain reaction (PCR) test
- COVID-19 negative: COVID-19 negative (i.e. no current or previous symptoms of COVID-19, confirmed PCR negative for COVID-19)
  Interventions: Diagnostic Test: SG Diagnostics COVID-19 Antigen Rapid Test Kit; Diagnostic Test: Polymerase chain reaction (PCR) test

INTERVENTIONS:
Diagnostic Test: SG Diagnostics COVID-19 Antigen Rapid Test Kit — SG Diagnostics COVID-19 Antigen Rapid Test Kit (self-use)
Diagnostic Test: Polymerase chain reaction (PCR) test — Professional collection of a second swab sample, for confirmation by PCR

SUMMARY:
The SG Diagnostics COVID-19 Antigen Rapid Test Kit (Colloidal Gold-Based) is a single-use test kit intended to detect the novel coronavirus SARS-CoV-2 that causes COVID-19. This test is intended for use with self-collected nasal swab samples in individuals who are suspected of COVID-19. This test utilizes a lateral flow immunoassay technology for the qualitative detection of spike and nucleocapsid protein antigens of SARS-CoV-2 in individuals with known or suspected COVID-19.

ELIGIBILITY:
Inclusion Criteria:

* Adult (aged ≥ 18 years) volunteers

Exclusion Criteria:

* Children (aged < 18years)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Volunteers with or without COVID-19 symptoms
Sampling Method: Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2021-05-11 (Actual); Primary Completion 2021-06-30 (Estimated); Study Completion 2021-07-10 (Estimated)

PRIMARY OUTCOMES:
Sensitivity of SG Diagnostics COVID-19 Antigen Rapid Test Kit | within 1 day
  Sensitivity of SG Diagnostics COVID-19 Antigen Rapid Test Kit (self-use)
Specificity of SG Diagnostics COVID-19 Antigen Rapid Test Kit | within 1 day
  Specificity of SG Diagnostics COVID-19 Antigen Rapid Test Kit (self-use)

CONTACTS AND LOCATIONS:
Locations (1):
- Maria Sklodowska-Curie Medical Academy, Warsaw, Poland

IPD SHARING:
Plan to Share IPD: Undecided